CLINICAL TRIAL: NCT00491764
Title: An Investigator-Blinded Study Evaluating the Efficacy and Safety of Four Posaconazole Treatment Regimens With Placebo and Terbinafine in the Treatment of Onychomycosis of the Toenail
Brief Title: A Study to Evaluate Efficacy and Safety of Four Posaconazole Regimens With Placebo and Terbinafine in the Treatment of Toenail Onychomycosis (Study P05082AM2)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05082
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — posaconazole; Terbinafine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Posaconazole 100 mg QD for 24 weeks. (Experimental): Posaconazole oral suspension (40 mg/mL) 100 mg QD for 24 weeks.
  Interventions: Drug: SCH 56592
- Posaconazole 200 mg QD for 24 weeks. (Experimental): Posaconazole oral suspension (40 mg/mL) 200 mg QD for 24 weeks.
  Interventions: Drug: SCH 56592
- Posaconazole 400 mg QD for 24 weeks. (Experimental): Posaconazole oral suspension (40 mg/mL) 400 mg QD for 24 weeks.
  Interventions: Drug: SCH 56592
- Posaconazole 400 mg QD for 12 weeks. (Experimental): Posaconazole oral suspension (40 mg/mL) 400 mg QD for 12 weeks.
  Interventions: Drug: SCH 56592
- Terbinafine (Active Comparator): Terbinafine 250 mg QD for 12 weeks.
  Interventions: Drug: Terbinafine
- Placebo (Placebo Comparator): Placebo for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 56592 — Posaconazole oral suspension (40 mg/mL) 100 mg QD for 24 weeks.
  Other Names: Posaconazole; Noxafil
  Arms: Posaconazole 100 mg QD for 24 weeks.
Drug: SCH 56592 — Posaconazole oral suspension (40 mg/mL) 200 mg QD for 24 weeks.
  Other Names: Posaconazole; Noxafil
  Arms: Posaconazole 200 mg QD for 24 weeks.
Drug: SCH 56592 — Posaconazole oral suspension (40 mg/mL) 400 mg QD for 24 weeks.
  Other Names: Posaconazole; Noxafil
  Arms: Posaconazole 400 mg QD for 24 weeks.
Drug: SCH 56592 — Posaconazole oral suspension (40 mg/mL) 400 mg QD for 12 weeks.
  Other Names: Posaconazole; Noxafil
  Arms: Posaconazole 400 mg QD for 12 weeks.
Drug: Terbinafine — Terbinafine 250 mg QD for 12 weeks.
  Arms: Terbinafine
Drug: Placebo — Placebo for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of oral administration of four dosing regimens of posaconazole relative to placebo and terbinafine, in the treatment of toenail onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet ALL the criteria listed below for entry:

  * Subject must be between 18 and 75 years of age inclusive, of either sex, and of any race;
  * Subject must have distal subungual infection that affects approximately 25% to 75% of at least one great toenail, both clinically and mycologically diagnosed;
  * Subject must have at least 2 mm of the proximal end of the target toenail free of infection;
  * Subject must have a target toenail that is assessed as capable of growing approximately 1 mm/month, (eg, the subject needs to report cutting his or her toenails at least once per month);
  * Subject must have liver function tests within 1.5 x the upper limit of normal (bilirubin and transaminases);
  * Subject must have normal serum creatinine levels;
  * Subject must be able to take study medication orally;
  * Subject must have no history of current narcotic or alcohol addiction;
  * Subject must be willing to give written informed consent and able to adhere to dose, procedures, and visit schedules;
  * Woman of childbearing potential who is currently sexually active must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 30 days after stopping the medication. Methods include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, oral or systemic hormonal contraceptive (plus an additional reliable barrier method), and surgical sterilization (eg, hysterectomy or tubal ligation).

Woman of child-bearing potential who is not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.

* Woman of childbearing potential must have a negative serum pregnancy test within 72 hours prior to start of study drug.

Exclusion Criteria:

* The subject will be excluded from entry if ANY of the criteria listed below are met:

  * Subject with one or more of the following conditions on the target toenail:

    * proximal subungual onychomycosis,
    * white superficial onychomycosis,
    * dermatophytoma or "yellow spike/streak",
    * exclusively lateral disease,
    * inability to become normal in the opinion of the investigator.
  * Subject with psoriasis, severe moccasin-type tinea pedis requiring treatment, symptomatic interdigital tinea pedis, lichen planus, or other abnormalities that could result in a clinically abnormal nail;
  * Subject with peripheral vascular disease or peripheral circulatory impairment;
  * Subject with history of uncontrolled diabetes mellitus;
  * Subject with known chronic or active liver disease;
  * Subject with any known immunodeficiency;
  * Subject with a family history of long QT syndrome;
  * Subject with an electrocardiogram with QTc interval prolongation greater than 450 msec for males and 470 msec for females;
  * Subject with potassium or magnesium lower than the lower limit of normal;
  * Subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study;
  * Subject who has received systemic antifungal therapy within 3 months or topical antifungal therapy applied to the foot or toenails within 1 month of study entry;
  * Subject who has received radiation therapy, chemotherapy, and/or immunosuppressive drugs within 6 months of Randomization, and/or oral corticosteroids for >1 month within the 6 months of Randomization (exception: inhaled steroids);
  * Subject using medications known to interact with azoles such as terfenadine, pimozide, quinidine, halofantrine, astemizole, alfentanil, cisapride, HMG-Co A (3-hydroxy-3-methylglutaryl coenzyme A) reductase inhibitors that are metabolized by CYP3A4, and ebastine, within 7 days prior to Randomization; and pravastatin within 14 days prior to Randomization;
  * Subject using medications known to lower the serum concentration/efficacy of azoles including rifampin, rifabutin, cimetidine, carbamazepine, phenytoin, barbiturates, and isoniazid, 3 doses or more within 7 days prior to Randomization;
  * Subject with a known sensitivity to azoles, POS and/or its excipients, terbinafine and/or its excipients;
  * Subject who has been previously enrolled in this study or any other POS investigational trial;
  * Subject known to have received treatment with investigational drugs within 30 days prior to enrollment into this study;
  * Woman who is breastfeeding, pregnant, or intends to become pregnant;
  * Subject who is part of the staff personnel directly involved with this study;
  * Subject who is a family member of the investigational study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Elewski B, Pollak R, Ashton S, Rich P, Schlessinger J, Tavakkol A. A randomized, placebo- and active-controlled, parallel-group, multicentre, investigator-blinded study of four treatment regimens of posaconazole in adults with toenail onychomycosis. Br J Dermatol. 2012 Feb;166(2):389-98. doi: 10.1111/j.1365-2133.2011.10660.x. Epub 2011 Dec 6. PMID 21967490

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 690 subjects were enrolled in the study and screened for eligibility. A total of 472 were screen-failures, leaving 218 subjects randomized to treatment.
Groups:
- Posaconazole 100 mg QD for 24 Weeks: Posaconazole oral suspension (40 mg/mL) 100 mg daily (QD) for 24 weeks.
- Terbinafine 250 mg QD for 12 Weeks.: Terbinafine 250 mg QD for 12 weeks.
- Placebo for 24 Weeks: Placebo for 24 weeks.
Period: Overall Study
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 12 Weeks. | Terbinafine 250 mg QD for 12 Weeks. | Placebo for 24 Weeks
Started | 37 | 37 | 36 | 36 | 36 | 36
Completed | 32 | 30 | 28 | 28 | 33 | 27
Not Completed | 5 | 7 | 8 | 8 | 3 | 9
Not completed — Adverse Event | 1 | 2 | 4 | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 2 | 2 | 4
Not completed — Non Compliance with the Protocol | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not Meet Protocol Eligibility | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Administrative | 1 | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 12 Weeks. | Terbinafine 250 mg QD for 12 Weeks. | Placebo for 24 Weeks | Total
Number analyzed (Participants) | 37 | 37 | 36 | 36 | 36 | 36 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.0) | 53.6 (10.8) | 49.9 (13.2) | 53.5 (11.8) | 50.1 (12.2) | 48.4 (14.8) | 50.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 8 | 7 | 7 | 7 | 45
  Male | 27 | 31 | 28 | 29 | 29 | 29 | 173

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure of Onychomycosis at Week 48.
Description: Complete cure is defined as negative mycology (negative culture and KOH [potassium hydroxide]) and 0% nail involvement (defined as absence of onycholysis and subungual hyperkeratosis).
Time Frame: Measured at Day 1, Week 2, Week 4, and Every 4 Weeks Thereafter Until Week 48
Population: This analysis was based on all randomized subjects who had a baseline assessment and at least one post-baseline assessment available, and who had been exposed to at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 12 Weeks. | Terbinafine 250 mg QD for 12 Weeks. | Placebo for 24 Weeks
Number analyzed (Participants) | 35 | 37 | 33 | 35 | 35 | 32
Participants | 8 | 20 | 15 | 7 | 13 | 0
Statistical Analysis 1: Comparison: Posaconazole 100 mg QD for 24 Weeks vs Placebo for 24 Weeks; Test type: Superiority or Other; p = 0.005, Fisher Exact; Mean Difference (Net) = 22.9, 95% CI [8.9 to 36.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 2: Comparison: Posaconazole 200 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 54.1, 95% CI [38.0 to 70.1] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 3: Comparison: Posaconazole 400 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 45.5, 95% CI [28.5 to 62.4] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 4: Comparison: Posaconazole 400 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p = 0.012, Fisher Exact; Mean Difference (Net) = 20.0, 95% CI [6.7 to 33.3] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 5: Comparison: Terbinafine 250 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 37.1, 95% CI [21.1 to 53.2] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions

2. Secondary Outcome: Effective Treatment of Onychomycosis at Week 48.
Description: Effective treatment is defined as negative mycology (negative culture and KOH) and either 0% nail involvement or >5 mm growth of unaffected nail
Time Frame: Measured at Day 1, Week 2, Week 4, and Every 4 Weeks Thereafter Until Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 12 Weeks. | Terbinafine 250 mg QD for 12 Weeks. | Placebo for 24 Weeks
Number analyzed (Participants) | 35 | 37 | 33 | 35 | 35 | 32
Participants | 9 | 24 | 16 | 11 | 19 | 0
Statistical Analysis 1: Comparison: Posaconazole 100 mg QD for 24 Weeks vs Placebo for 24 Weeks; Test type: Superiority or Other; p = 0.002, Fisher Exact; Mean Difference (Net) = 25.7, 95% CI [11.2 to 40.2] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 2: Comparison: Posaconazole 200 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 64.9, 95% CI [49.5 to 80.2] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 3: Comparison: Posaconazole 400 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 48.5, 95% CI [31.4 to 65.5] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 4: Comparison: Posaconazole 400 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 31.4, 95% CI [16.0 to 46.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 5: Comparison: Terbinafine 250 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 54.3, 95% CI [37.8 to 70.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions

3. Secondary Outcome: Treatment Success of Onychomycosis at Week 48
Description: Treatment success was defined as negative mycology (negative culture and negative KOH) and =<10% nail involvement.
Time Frame: Measured at Day 1, Week 2, Week 4, and Every 4 Weeks Thereafter Until Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 24 Weeks. | Posaconazole 400 mg QD for 12 Weeks. | Terbinafine 250 mg QD for 12 Weeks. | Placebo for 24 Weeks
Number analyzed (Participants) | 35 | 37 | 33 | 35 | 35 | 32
Participants | 11 | 24 | 22 | 11 | 20 | 0
Statistical Analysis 1: Comparison: Posaconazole 100 mg QD for 24 Weeks vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 31.4, 95% CI [16.0 to 46.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 2: Comparison: Posaconazole 200 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 64.9, 95% CI [49.5 to 80.2] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 3: Comparison: Posaconazole 400 mg QD for 24 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 66.7, 95% CI [50.6 to 82.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 4: Comparison: Posaconazole 400 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 31.4, 95% CI [16.0 to 46.8] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions
Statistical Analysis 5: Comparison: Terbinafine 250 mg QD for 12 Weeks. vs Placebo for 24 Weeks; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 57.1, 95% CI [40.7 to 73.5] — Difference is in the proportion for Yes responders. Confidence Interval is around the difference in proportions

ADVERSE EVENTS:
Description: Number of participants at risk included the 216 subjects who received treatment. Of the 218 subjects randomized, 1 subject in the posaconazole 100 mg and 1 subject in the placebo group were not treated.
Arm/Group | Posaconazole 100 mg QD for 24 Weeks | Posaconazole 200 mg QD for 24 Weeks | Posaconazole 400 mg QD for 24 Weeks | Posaconazole 400 mg QD for 12 Weeks | Terbinafine 250 mg QD for 12 Weeks | Placebo for 24 Weeks
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/37 | 1/36 | 1/36 | 0/36 | 3/35
Other Adverse Events (participants affected / at risk) | 26/36 | 21/37 | 20/36 | 18/36 | 20/36 | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole 100 mg QD for 24 Weeks (N=36) | Posaconazole 200 mg QD for 24 Weeks (N=37) | Posaconazole 400 mg QD for 24 Weeks (N=36) | Posaconazole 400 mg QD for 12 Weeks (N=36) | Terbinafine 250 mg QD for 12 Weeks (N=36) | Placebo for 24 Weeks (N=35)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole 100 mg QD for 24 Weeks (N=36) | Posaconazole 200 mg QD for 24 Weeks (N=37) | Posaconazole 400 mg QD for 24 Weeks (N=36) | Posaconazole 400 mg QD for 12 Weeks (N=36) | Terbinafine 250 mg QD for 12 Weeks (N=36) | Placebo for 24 Weeks (N=35)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (7) | 1 (1) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (6) | 0 (0) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (6) | 2 (2) | 1 (4) | 0 (0) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
PAIN (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SEASONAL ALLERGY (Immune system disorders) | 2 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
INFLUENZA (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
LARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 4 (6) | 3 (3) | 6 (7) | 2 (4) | 3 (3) | 6 (6)
SINUSITIS (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
TINEA PEDIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 1 (1) | 3 (3) | 6 (7) | 5 (5) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 1 (1) | 1 (13) | 3 (3) | 3 (3) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 4 (5) | 2 (3) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
ONYCHALGIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide to sponsor 45 days prior to submission for publication/presentation, review copies of content to be presented that contains any results of the study. The sponsor has the right to review/comment with regard to proprietary information, accuracy, and fair balance. If disagreements arise concerning appropriateness of content to be presented, investigator must meet with sponsor prior to submission for publication to make good faith efforts to discuss/resolve any issues/disagreement.